CLINICAL TRIAL: NCT06426043
Title: An Exploratory Study on the Efficacy and Safety of Lusutrombopag in the Treatment of Recurrent/Refractory/Intolerable NSAA
Brief Title: A Prospective Study on the Treatment of Recurrent/Refractory/Intolerable NSAA With Lusutrombopag
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNA-2024
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Aplastic Anemia
Keywords: Non-severe aplastic anemia; Lusutrombopag; Refractory; Recurrent
MeSH Terms: conditions — Anemia, Aplastic; Recurrence | interventions — lusutrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lusutrombopag (Experimental): Administer lusutrombopag at 3mg/qd orally for 12 weeks (lusutrombopag starting dose is 3mg, once daily. After 2 weeks of continuous administration, the dose can be increased by 3mg every 2 weeks based on the platelet count and safety of the subject. The dose can be gradually increased to 9mg/d over a total of 12 weeks). The course should be at least 3 months. When the platelet increase is <20×10^9/L, the daily dose can be increased by 3mg up to a maximum of 9mg/day; when the platelet increase is ≥50×10^9/L and ≤200×10^9/L, the dose can be maintained; when the platelet count is ≥200×10^9/L and ≤400×10^9/L, the daily dose can be reduced by 3mg; when the platelet count is >400×10^9/L, the drug can be suspended and resumed when the platelet count decreases to <200×10^9/L, with the daily dose reduced by 3mg. In this case, if the lowest dose of 3mg/day is used, the drug can be suspended. Responders continue treatment until 6 months.
  Interventions: Drug: Lusutrombopag

INTERVENTIONS:
Drug: Lusutrombopag — Administer lusutrombopag at 3mg/qd orally for 12 weeks (lusutrombopag starting dose is 3mg, once daily. After 2 weeks of continuous administration, the dose can be increased by 3mg every 2 weeks based on the platelet count and safety of the subject. The dose can be gradually increased to 9mg/d over a total of 12 weeks). The course should be at least 3 months. When the platelet increase is <20×109/L, the daily dose can be increased by 3mg up to a maximum of 9mg/day; when the platelet increase is ≥50×10^9/L and ≤200×10^9/L, the dose can be maintained; when the platelet count is ≥200×10^9/L and ≤400×10^9/L, the daily dose can be reduced by 3mg; when the platelet count is >400×10^9/L, the drug can be suspended and resumed when the platelet count decreases to <200×10^9/L, with the daily dose reduced by 3mg. In this case, if the lowest dose of 3mg/day is used, the drug can be suspended. Responders continue treatment until 6 months.

SUMMARY:
In a prospective, single-arm study, the efficacy and safety of Lusutrombopag in the treatment of relapsed/refractory/intolerable non-severe aplastic anemia (NSAA) were explored.

DETAILED DESCRIPTION:
The enrolled patients: were given Lusutrombopag at 3mg/qd orally for 12 weeks (the starting dose of lusutrombopag was 3mg, taken once daily. After 2 weeks of continuous administration, the dose was increased by 3mg every 2 weeks based on the platelet count and safety of the subjects. The dose was gradually increased to 9mg/d over a total of 12 weeks). The treatment duration was at least 3 months. When the platelet increase was <20×10^9/L, the daily dose was increased by 3mg, up to a maximum of 9mg/day. When the platelet increase was ≥50×109/L and ≤200×10^9/L, the dose was maintained at the previous level. When the platelet count was ≥200×10^9/L and ≤400×10^9/L, the daily dose was reduced by 3mg. When the platelet count was >400×10^9/L, the drug could be suspended, and the dose was reduced by 3mg when the platelet count decreased to <200×10^9/L. In this case, if the lowest dose of 3mg/day was used, the drug could be suspended. Responders continued treatment for 6 months. Other TPO-RA therapies were not allowed during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years old, male or female.
2. Participants must be diagnosed with NSAA and have a refractory/relapsed/intolerable response to standard-dose cyclosporine (CsA). The definition of refractory/relapsed is patients who have been treated with sufficient doses of cyclosporine (3-5mg/kg) for at least 6 months without response or relapse. The definition of intolerable is patients who cannot tolerate CsA and have stopped treatment due to significant side effects.
3. Participants must meet the following criteria at enrollment: platelets <30×109/L.
4. Baseline liver and kidney function must be within 2 times of normal range.
5. No active infection; no pregnancy or breastfeeding.
6. Participants must agree to sign the informed consent form.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.

Exclusion Criteria:

1. Other causes of pancytopenia, such as myelodysplastic syndrome (MDS).
2. Evidence of clonal hematopoietic system bone marrow disease (MDS, AML) with cytogenetics.
3. PNH clone ≥50%.
4. Received hematopoietic stem cell transplant (HSCT) prior to enrollment.
5. Received ATG treatment within 6 months prior to enrollment.
6. Infection or bleeding that cannot be controlled with standard therapy.
7. Allergic to ruxolitinib.
8. Active HIV, HCV, or HBV infection, cirrhosis, or portal hypertension.
9. Any malignant tumor within 5 years, or local basal cell carcinoma of the skin.
10. History of thromboembolic events, myocardial infarction, or stroke (including antiphospholipid syndrome) and current use of anticoagulants.
11. Pregnant or breastfeeding (lactating) women.
12. Participated in another clinical trial within 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate at 3 months | 3 month
  Proportion of patients who achieved complete response, partial response and hematological response
Overall response rate at 6 months | 6 month
  Proportion of patients who achieved complete response, partial response and hematological response

SECONDARY OUTCOMES:
adverse event rate at 3 months | 3 month
  Proportion of patients with adverse eventsProportion of patients with adverse events
adverse event rate at 6 months | 6 month
  Proportion of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bing Bing, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young NS. Aplastic Anemia. N Engl J Med. 2018 Oct 25;379(17):1643-1656. doi: 10.1056/NEJMra1413485. No abstract available. PMID 30354958
- [Background] Ruan J, Zuo W, Chen M, Yang C, Han B. Eltrombopag is effective in patients with relapse/refractory aplastic anemia-report from a single center in China. Ann Hematol. 2020 Dec;99(12):2755-2761. doi: 10.1007/s00277-020-04266-1. Epub 2020 Sep 17. PMID 32944791
- [Background] Katsube T, Wajima T, Fukuhara T, Kano T. Effects of Food and Calcium Carbonate on the Pharmacokinetics of Lusutrombopag, a Novel Thrombopoietin Receptor Agonist. Clin Ther. 2019 Sep;41(9):1747-1754.e2. doi: 10.1016/j.clinthera.2019.06.004. Epub 2019 Jul 11. PMID 31303281
- [Background] Hidaka H, Kurosaki M, Tanaka H, Kudo M, Abiru S, Igura T, Ishikawa T, Seike M, Katsube T, Ochiai T, Kimura K, Fukuhara T, Kano T, Nagata T, Tanaka K, Kurokawa M, Yamamoto K, Osaki Y, Izumi N, Imawari M. Lusutrombopag Reduces Need for Platelet Transfusion in Patients With Thrombocytopenia Undergoing Invasive Procedures. Clin Gastroenterol Hepatol. 2019 May;17(6):1192-1200. doi: 10.1016/j.cgh.2018.11.047. Epub 2018 Nov 28. PMID 30502505
- [Background] Wan Z, Chen M, Han B. Avatrombopag, a promising novel thrombopoietin receptor agonist for refractory/relapsed/intolerant non-severe aplastic anemia: a phase 2 single-arm clinical trial. Ann Med. 2023 Dec;55(1):2224044. doi: 10.1080/07853890.2023.2224044. PMID 37318085